CLINICAL TRIAL: NCT06413381
Title: Risk Factors for Non-response to Hormonal Medical Therapy in Patients With Endometriosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOFAIL - 01
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-03

CONDITIONS: Endometriosis
Keywords: pelvic pain; endometriosis; hormone therapy; therapeutic non-response; risk factors; reproduction; infertility
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus group: non-responsive patients to medical treatment
- Control group: responsive patients to medical treatment

SUMMARY:
Determine the proportion of patients with endometriosis unresponsive to medical therapy and to compare the clinical and ultrasonographic characteristics of this group of patients (study group) with the clinical and ultrasonographic characteristics of patients responsive to medical therapy (control group).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years;
* patients with endometriosis-related pain symptoms (dyspareunia, dyschezia, dysmenorrhea, chronic pelvic pain, dysuria, periovulatory pain, with at least one of these symptoms presenting Numerical Pain Rating Scale intensity > 5);
* indication for administration of oral hormonal medical treatment for endometriosis;
* acquisition of informed consent.

Exclusion Criteria:

* patients with contraindications to oral hormone treatment
* current or previous pelvic infections
* history of malignancy or current suspicion of gynecologic malignant lesions
* previous pelvic surgery (hysterectomy, salpingectomy, ovarian cyst removal, myomectomy, surgery for endometriosis, bowel resections)
* positive history of other causes of chronic pelvic pain
* post-menopausal status

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with clinical and ultrasound diagnosis of endometriosis with indication for administration of hormone therapy
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with endometriosis non-responsive to medical treatment at 12 months | 12 months
  determine the rate of patients with endometriosis who were non-responsive to medical treatment at 12 months and to compare the clinical and ultrasound characteristics of this group of patients (study group) with the clinical and ultrasound characteristics of patients responsive to medical treatment (control group).

SECONDARY OUTCOMES:
Rate of patients with endometriosis non-responsive to medical treatment at 6 months | 6 months
  determine the rate of patients with endometriosis who were non-responsive to medical treatment at 6 months and to compare the clinical and ultrasound characteristics of this group of patients (study group) with the clinical and ultrasound characteristics of patients responsive to medical treatment (control group).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria, Policlinico Sant'Orsola, Bologna, BO, Italy